CLINICAL TRIAL: NCT00552487
Title: Isolated ACTH Deficiency in Patients With Hashimoto Thyroiditis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wuerzburg (Other)
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 112/05
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Hashimoto Disease; Adrenal Insufficiency
Keywords: isolated ACTH deficiency; Hashimoto disease; Hashimoto thyroiditis; autoimmune thyroiditis
MeSH Terms: conditions — Hashimoto Disease; Adrenal Insufficiency; ACTH Deficiency, Isolated; Thyroiditis, Autoimmune | interventions — adrenocorticotropin zinc; Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Other): healthy people without Hashimoto disease receive a 1µg ACTH stimulation test
  Interventions: Drug: synacthen
- 2 (Other): patients with Hashimoto disease with well being receive a 1 µg ACTH stimulation test
  Interventions: Drug: synacthen
- 3 (Other): patients with Hashimoto disease an impaired well-being receive a 1 µg ACTH stimulation test
  Interventions: Drug: synacthen
- 4 (Other): patients with Hashimoto disease and negative TPO antibodies receive a 1µg ACTH stimulation test
  Interventions: Drug: synacthen

INTERVENTIONS:
Drug: synacthen — 1 µg synacthen in the vein
  Other Names: ACTH

SUMMARY:
The purpose of this study is to determine whether patients with Hashimoto thyroiditis and impaired well-being may have a partial secondary adrenocortical insufficiency.

DETAILED DESCRIPTION:
Many patients with Hashimoto thyroiditis who are correctly substituted with thyroid hormones have an impaired well-being. in some people an isolated ACTH deficiency was found.

In this study a 1 µg ACTH test is performed to evaluate the adrenocortical function.

ELIGIBILITY:
Inclusion Criteria:

* Hashimoto thyroiditis euthyreot thyroid function with levothyroxin therapy written informed consent

Exclusion Criteria:

* • hypothyroidism of other origin

  * pregnancy and lactation
  * oral contraception
  * glucocorticoid therapy during the last 2 months
  * History of malignancy or chronic infections (Hepatitis, HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-10; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
serum cortisol-peak 30 min after ACTH-stimulation | 30 minutes

SECONDARY OUTCOMES:
serum DHEA-peak 30 min. after ACTH-stimulation,DHEA-S, ACTH | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Allolio, MD, Principal Investigator — University of Wuerzburg
Locations (1):
- University of Wuerzburg, Department of Endocrinology, Würzburg, Bavaria, Germany